CLINICAL TRIAL: NCT05356273
Title: The Effect of Massage on the Bilirubin Level in Term Infants Receiving Phototherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/84
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2022-09

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: infant; baby massage; hyperbilirubinemia; bilirubin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Massage Group (Experimental): The incubator temperature was adjusted between 28-30 C, and it was administered while the baby was awake and one hour after feeding. Before the massage, the hands were washed and warmed. Just before each phototherapy application, 10-minute baby massage was performed by the researcher.Then phototherapy was applied.
  Interventions: Procedure: Baby massage
- Control Group (No Intervention): Just received phototherapy twice a day

INTERVENTIONS:
Procedure: Baby massage — Starting from the baby's face first, then the abdomen and chest, back, upper extremities and finally the lower extremities were massaged with semi-circular movements, respectively.
  Arms: Massage Group

SUMMARY:
Background: It has been reported in the current literature that massage has various positive physiological effects on the newborn. Also baby massage; It increases the collection and excretion of waste products such as bilirubin by accelerating the flow of blood, lymph and tissue fluids. Our aim is to investigate the effect of infant massage on hyperbilirubinemia in newborns receiving phototherapy.

Method: The population of the study consisted of babies who were hospitalized in Istanbul Haseki Training and Research Hospital Neonatal Intensive Care Unit between October 2021 and January 2022 and needed phototherapy. Transcutaneous bilirubin device and data collection form were used to obtain the data. 61 newborns who met the study criteria were randomly divided into experimental (n=30) and control (n=31) groups. Phototherapy was applied to all babies twice a day. In addition to phototherapy, infant massage was applied to the experimental group for 10 minutes just before the phototherapy. Bilirubin level measurements were made 2 hours after the end of phototherapy for both groups. Diaper changes for both groups were carried out 8 times a day, every 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* Born between 37-42 gestational weeks
* Birth weight between 2500-4000gr
* 1st and 5th Apgar score between 7-10
* Needing phototherapy treatment
* Diagnosed with indirect hyperbilirubinemia 24 hours or more after birth
* Orally fed
* No health problems other than indirect hyperbilirubinemia
* Newborns who has stable vital signs

Exclusion Criteria:

* ABO blood incompatibility or Rh incompatibility
* Diagnosed with direct hyperbilirubinemia
* Newborns who has skin anomaly
* Needing fluid replacement
* Newborns with gastrointestinal disorders

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Bilirubin levels | 72 hours
  decreasing bilirubin levels within intervention times

SECONDARY OUTCOMES:
Stool frequency | 72 hours
  increasing stool frequency within intervention times

CONTACTS AND LOCATIONS:
Overall Officials: Elif Dogan, Principal Investigator — Researcher Assistant
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmadipour S, Mardani M, Mohsenzadeh A, Baharvand P, Nazeri MG. The Lowering of Bilirubin Levels in Full-Term Newborns by the Effect of Combined Massage Therapy and Phototherapy Practice. Am J Perinatol. 2024 May;41(S 01):e3420-e3424. doi: 10.1055/s-0039-1685493. Epub 2019 Apr 18. PMID 30999382
- [Background] Amos RC, Jacob H, Leith W. Jaundice in newborn babies under 28 days: NICE guideline 2016 (CG98). Arch Dis Child Educ Pract Ed. 2017 Aug;102(4):207-209. doi: 10.1136/archdischild-2016-311556. Epub 2017 Feb 8. No abstract available. PMID 28179382
- [Background] Anderson NB, Calkins KL. Neonatal Indirect Hyperbilirubinemia. Neoreviews. 2020 Nov;21(11):e749-e760. doi: 10.1542/neo.21-11-e749. PMID 33139512
- [Background] Basiri-Moghadam M, Basiri-Moghadam K, Kianmehr M, Jani S. The effect of massage on neonatal jaundice in stable preterm newborn infants: a randomized controlled trial. J Pak Med Assoc. 2015 Jun;65(6):602-6. PMID 26060154
- [Background] Dalili H, Sheikhi S, Shariat M, Haghnazarian E. Effects of baby massage on neonatal jaundice in healthy Iranian infants: A pilot study. Infant Behav Dev. 2016 Feb;42:22-6. doi: 10.1016/j.infbeh.2015.10.009. Epub 2015 Nov 29. PMID 26646074
- [Background] Eghbalian F, Rafienezhad H, Farmal J. The lowering of bilirubin levels in patients with neonatal jaundice using massage therapy: A randomized, double-blind clinical trial. Infant Behav Dev. 2017 Nov;49:31-36. doi: 10.1016/j.infbeh.2017.05.002. Epub 2017 Jul 6. PMID 28688960
- [Background] Garg BD, Kabra NS, Balasubramanian H. Role of massage therapy on reduction of neonatal hyperbilirubinemia in term and preterm neonates: a review of clinical trials. J Matern Fetal Neonatal Med. 2019 Jan;32(2):301-309. doi: 10.1080/14767058.2017.1376316. Epub 2017 Sep 13. PMID 28870134
- [Background] Gozen D, Yilmaz OE, Dur S, Caglayan S, Tastekin A. Transcutaneous bilirubin levels of newborn infants performed abdominal massage: A randomized controlled trial. J Spec Pediatr Nurs. 2019 Apr;24(2):e12237. doi: 10.1111/jspn.12237. Epub 2019 Feb 28. PMID 30817090
- [Background] Korkmaz G, Esenay FI. Effects of Massage Therapy on Indirect Hyperbilirubinemia in Newborns Who Receive Phototherapy. J Obstet Gynecol Neonatal Nurs. 2020 Jan;49(1):91-100. doi: 10.1016/j.jogn.2019.11.004. Epub 2019 Dec 6. PMID 31812490
- [Background] Lei M, Liu T, Li Y, Liu Y, Meng L, Jin C. Effects of massage on newborn infants with jaundice: A meta-analysis. Int J Nurs Sci. 2018 Jan 31;5(1):89-97. doi: 10.1016/j.ijnss.2018.01.004. eCollection 2018 Jan 10. PMID 31406807
- [Background] Lin CH, Yang HC, Cheng CS, Yen CE. Effects of infant massage on jaundiced neonates undergoing phototherapy. Ital J Pediatr. 2015 Nov 25;41:94. doi: 10.1186/s13052-015-0202-y. PMID 26607061
- [Background] Lori Kenari R, Aziznejadroshan P, Haghshenas Mojaveri M, Hajian-Tilaki K. Comparing the effect of kangaroo mother care and field massage on serum bilirubin level of term neonates with hyperbilirubinemia under phototherapy in the neonatal ward. Caspian J Intern Med. 2020 Winter;11(1):34-40. doi: 10.22088/cjim.11.1.34. PMID 32042384
- [Background] Mitra S, Rennie J. Neonatal jaundice: aetiology, diagnosis and treatment. Br J Hosp Med (Lond). 2017 Dec 2;78(12):699-704. doi: 10.12968/hmed.2017.78.12.699. PMID 29240507
- [Background] Olusanya BO, Kaplan M, Hansen TWR. Neonatal hyperbilirubinaemia: a global perspective. Lancet Child Adolesc Health. 2018 Aug;2(8):610-620. doi: 10.1016/S2352-4642(18)30139-1. Epub 2018 Jun 28. PMID 30119720
- [Background] Pace EJ, Brown CM, DeGeorge KC. Neonatal hyperbilirubinemia: An evidence-based approach. J Fam Pract. 2019 Jan/Feb;68(1):E4-E11. PMID 30724909
- [Background] Zhang M, Wang L, Wang Y, Tang J. The influence of massage on neonatal hyperbilirubinemia: a meta-analysis of randomized controlled trials. J Matern Fetal Neonatal Med. 2019 Sep;32(18):3109-3114. doi: 10.1080/14767058.2018.1455183. Epub 2018 Apr 9. PMID 29631455
- [Background] Montgomery P, Grant S, Mayo-Wilson E, Macdonald G, Michie S, Hopewell S, Moher D; CONSORT-SPI Group. Reporting randomised trials of social and psychological interventions: the CONSORT-SPI 2018 Extension. Trials. 2018 Jul 31;19(1):407. doi: 10.1186/s13063-018-2733-1. PMID 30060754